CLINICAL TRIAL: NCT03356678
Title: Pralatrexate for Relapsed or Refractory Peripheral T-cell Lymphoma: a Multicenter, Multinational Retrospective Analysis
Brief Title: Pralatrexate for Relapsed or Refractory Peripheral T-cell Lymphoma
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Seog Kim, MD, Samsung Medical Center
Other Study IDs: 2016-09-090
Record Dates: First submitted 2017-07-19; First posted 2017-11-29 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Relapsed or Refractory Peripheral T-cell Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, T-Cell, Peripheral | interventions — 10-propargyl-10-deazaaminopterin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Pralatrexate — * Patients treated with pralatrexate due to relapse or refractory disease after primary and/or salvage treatment. Relapse following an autologous stem cell transplant allowed.
  * Patients treated with pralatrexate 30mg/m2 once a week for 6 weeks as part of a 7-week cycle. However, modified dose and/or schedule allowed.

SUMMARY:
A non-interventional, multicenter, multinational retrospective analysis using electronic case report forms completed by the investigators based on information from patient medical records

DETAILED DESCRIPTION:
All patients who satisfy the inclusion criteria for this study in each participating institution will be included. Considering the number of participating centers in Korea, Latin America (Mexico, Colombia), and Europe (Switzerland, Israel), the expected number of patients is 50.

This research involves only the collection and analysis of existing data, documents, and records. The information will be recorded by the investigators on a CRF in a way that the subjects cannot be identified directly or through identifiers linked to the subjects. Thus, this study should be reviewed and approved by the Institutional Review Board of each participating institute, and exemption from additional written informed consent should be applied.

1. Age, sex, nationality, ethnicity
2. Ann Arbor stage, disease involved sites, number of extranodal involvement, serum LDH concentration, ECOG performance status, presence of B symptoms, regional lymph node involvement, International Prognostic Index, bone marrow invasion at the time of pralatrexate treatment
3. Dose and schedule of pralatrexate, start date, last treatment date, other treatment modalities

ELIGIBILITY:
Inclusion Criteria:

- 1. Histologically confirmed peripheral T-cell lymphoma according to following inclusion criteria of subtypes according to the 2016 revision of the World Health Organization classification of lymphoid neoplasm

1. Adult T-cell leukemia/lymphoma
2. Angioimmunoblastic T-cell lymphoma
3. Anaplastic large cell lymphoma, ALK positive
4. Anaplastic large cell lymphoma, ALK negative
5. Peripheral T-cell lymphoma, NOS
6. Enteropathy-type intestinal lymphoma
7. Hepatosplenic T-cell lymphoma
8. Extranodal NK/T-cell lymphoma, nasal type
9. Subcutaneous panniculitis-like T-cell lymphoma
10. Transformed mycosis fungoides
11. Mycosis fungoides
12. Sézary syndrome
13. Primary cutaneous CD30+T-cell lymphoproliferative disorder (primary cutaneous anaplastic large cell lymphoma)
14. Primary cutaneous gamma-delta T-cell lymphoma 2. Age ≥ 18 years old 3. Patients treated with pralatrexate due to relapse or refractory disease after primary and/or salvage treatment. Relapse following an autologous stem cell transplant allowed.

4. Patients treated with pralatrexate 30mg/m2 once a week for 6 weeks as part of a 7-week cycle. However, modified dose and/or schedule allowed.

Exclusion Criteria:

* 1. Histologically confirmed peripheral T-cell lymphoma with following exclusion criteria of subtypes

  1. Aggressive NK-cell leukemia
  2. T-cell prolymphocytic leukemia
  3. T-cell large granular lymphocytic leukemia
  4. Primary cutaneous CD30+ T-cell lymphoproliferative disorders (lymphomatoid papulosis) 2. Patients with active/symptomatic central nervous system (CNS) involvement. 3. HIV-related lymphoma 4. Prior allogeneic stem cell transplant within 6 months. 5. Concurrent active or history of other malignancies. 6. Concurrent uncontrolled serious medical or psychiatric conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who satisfy the inclusion criteria for this study in each participating institution will be included. Considering the number of participating centers in Korea, Latin America (Mexico, Colombia), and Europe (Switzerland, Israel), the expected number of patients is 50.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2016-09-23 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) including complete remission (CR) and partial remission (PR) | This is a restrospective study. Data collection and analysis will be done for 6 months.
  retrospective analysis using electronic case report forms completed by the investigators based on information from patient medical records

SECONDARY OUTCOMES:
Progression-free survival (PFS) | This is a restrospective study. Data collection and analysis will be done for 6 months.
  retrospective analysis using electronic case report forms completed by the investigators based on information from patient medical records
Overall survival (OS) | This is a restrospective study. Data collection and analysis will be done for 6 months.
  retrospective analysis using electronic case report forms completed by the investigators based on information from patient medical records
Duration of response (DoR) | This is a restrospective study. Data collection and analysis will be done for 6 months.
  retrospective analysis using electronic case report forms completed by the investigators based on information from patient medical records
Toxicity | This is a restrospective study. Data collection and analysis will be done for 6 months.
  This study will investigate the number of participants with grade 3-4 neutropenia, grade 3-4 thrombocytopenia, grade 3-4 anemia and grade 4 febrile neutropenia according to CTCAE v4.0.
  This study will also investigate the number of participants with nausea, anorexia, constipation, diarrhea, peirpheral neuropathy, and skin rash that are related pralatrexate treatment according to CTCAE v4.0.
Tolerability | This is a restrospective study. Data collection and analysis will be done for 6 months.
  This study will investigate the dose intensity of pralatrexate based in information from patient medical records.

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Samsung Medical Center, Seoul, Seoul, Korea, Republic of
  - 81, Irwon-ro, Gangnam-gu, Seoul, Republic of Korea, Seoul

IPD SHARING:
Plan to Share IPD: Undecided